CLINICAL TRIAL: NCT06508814
Title: Pain With Differing Insufflation Pressures During Laparoscopic Hysterectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-09977-FB
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 12 mmHg Insufflation Pressure (Experimental): Participants received 12 mmHg of insufflation pressure during their laparoscopic hysterectomy.
  Interventions: Procedure: Lower Insufflation Pressure
- 15 mmHg Insufflation Pressure (Active Comparator): Participants received 15 mmHg of insufflation pressure during their laparoscopic hysterectomy.
  Interventions: Procedure: Standard Insufflation Pressure

INTERVENTIONS:
Procedure: Lower Insufflation Pressure — Participants underwent laparoscopic hysterectomy with an insufflation pressure that is lower than the standard insufflation pressure used in this type of surgery.
  Arms: 12 mmHg Insufflation Pressure
Procedure: Standard Insufflation Pressure — Participants underwent laparoscopic hysterectomy with a standard insufflation pressure.
  Arms: 15 mmHg Insufflation Pressure

SUMMARY:
The purpose of this study is to determine the effect of decreased insufflation pressure on postoperative pain, analgesic use, and surgical safety and feasibility for laparoscopic hysterectomy.

DETAILED DESCRIPTION:
This is a prospective, single-blinded, randomized clinical trial in which participants undergoing laparoscopic hysterectomy will be randomized in a 1:1 ratio to undergo surgery with peritoneal insufflation pressure set to 15 mmHg (standard) or 12 mmHg (comparison). Randomization was performed using computer-generated permuted blocks of four participants. All participants on the first postoperative day will be asked to rate their pain with a Visual Analog Scale (VAS). At a postoperative visit 2 weeks after surgery, all participants will be asked to complete the VAS again. The highest preoperative pain (up to 2 hours before surgery) and immediate postoperative pain, using the VAS, in the post anesthesia care unit (PACU) will be recorded. All participants will be planned for discharge from PACU. Age, body mass index, gynecologic diagnosis, medical history, and preoperative analgesia or opioid use will be extracted from the medical records by trained research staff and entered into a secure electronic database. Preoperative analgesia and opioid saw will be verified with active prescription records at the time of surgery. After surgery, analgesic doses, operative time, additional procedures performed, conversion to laparotomy or increased insufflation pressure, estimated blood loss, and length of stay will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 80
* BMI 55.0 or less
* Laparoscopic hysterectomy surgery planned

Exclusion Criteria:

* Women younger than 18 or older than 80 years of age
* BMI over 55.0
* Laparoscopic hysterectomy surgery not planned

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women who are biologically female
Enrollment: 100 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2025-06-10 (Estimated); Study Completion 2025-06-10 (Estimated)

PRIMARY OUTCOMES:
Pain on postoperative day 1 | 24 hours following surgery
  All participants will be asked to rate their pain using the Visual Analog Scale (VAS) approximately 24 hours after surgery completion. This scale ranges from 0 to 10, with 0 indicating no pain and 10 indicating worst possible pain.

SECONDARY OUTCOMES:
Preoperative pain | Within 2 hours before surgery
  All participants will be asked to rate their pain using the Visual Analog Scale (VAS) upon their arrival before surgery. This scale ranges from 0 to 10, with 0 indicating no pain and 10 indicating worst possible pain.
Postoperative pain while in PACU | Approximately 2 hours after surgery completion
  All participants will be asked to rate their pain using the Visual Analog Scale (VAS) while they are recovering in PACU, approximately 2 hours after surgery completion. This scale ranges from 0 to 10, with 0 indicating no pain and 10 indicating worst possible pain.
Postoperative pain at follow-up visit | Approximately 2 weeks after surgery completion
  All participants will be asked to rate their pain using the Visual Analog Scale (VAS) at their 2-week postoperative follow-up visit. This scale ranges from 0 to 10, with 0 indicating no pain and 10 indicating worst possible pain.
Opioid use after discharge | Within 2 weeks after surgery
  All participants will be asked about the number of prescription opioid pills they took following discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tennessee Health Science Center, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rustia GM, Baracy MG Jr, Khair E, Hagglund KH, Aslam MF. Pain With Differing Insufflation Pressures During Robotic Sacrocolpopexy: A Randomized Controlled Trial. Obstet Gynecol. 2023 Jul 1;142(1):151-159. doi: 10.1097/AOG.0000000000005231. Epub 2023 Jun 7. PMID 37348093
- [Background] Song T, Kim KH, Lee KW. The Intensity of Postlaparoscopic Shoulder Pain Is Positively Correlated with the Amount of Residual Pneumoperitoneum. J Minim Invasive Gynecol. 2017 Sep-Oct;24(6):984-989.e1. doi: 10.1016/j.jmig.2017.06.002. Epub 2017 Jun 7. PMID 28602786
- [Background] Kyle EB, Maheux-Lacroix S, Boutin A, Laberge PY, Lemyre M. Low vs Standard Pressures in Gynecologic Laparoscopy: a Systematic Review. JSLS. 2016 Jan-Mar;20(1):e2015.00113. doi: 10.4293/JSLS.2015.00113. PMID 26955258
- [Background] Grant A, Keltz J, Huang K. Is Decreased Insufflation Pressure During Major Robotic-Assisted Gynecologic Surgery Associated With Decreased Recovery Time and Patient Reported Pain Score. J Minim Invasive Gynecol. 2015 Nov-Dec;22(6S):S26. doi: 10.1016/j.jmig.2015.08.075. Epub 2015 Oct 15. No abstract available. PMID 27679192
- [Background] Topcu HO, Cavkaytar S, Kokanali K, Guzel AI, Islimye M, Doganay M. A prospective randomized trial of postoperative pain following different insufflation pressures during gynecologic laparoscopy. Eur J Obstet Gynecol Reprod Biol. 2014 Nov;182:81-5. doi: 10.1016/j.ejogrb.2014.09.003. Epub 2014 Sep 16. PMID 25265495
- [Background] Angioli R, Terranova C, Plotti F, Cafa EV, Gennari P, Ricciardi R, Aloisi A, Miranda A, Montera R, De Cicco Nardone C. Influence of pneumoperitoneum pressure on surgical field during robotic and laparoscopic surgery: a comparative study. Arch Gynecol Obstet. 2015 Apr;291(4):865-8. doi: 10.1007/s00404-014-3494-z. Epub 2014 Sep 27. PMID 25260990

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-12): https://cdn.clinicaltrials.gov/large-docs/14/NCT06508814/Prot_SAP_000.pdf
  • Informed Consent Form (2024-05-31): https://cdn.clinicaltrials.gov/large-docs/14/NCT06508814/ICF_001.pdf